CLINICAL TRIAL: NCT01553981
Title: A Double Blind Randomized Control Trial of Tadalafil in Interstitial Lung Disease of Scleroderma
Brief Title: A Trial of Tadalafil in Interstitial Lung Disease of Scleroderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Vikas Agarwal, Additional Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGI/BE/06/2012
Record Dates: First submitted 2012-03-11; First posted 2012-03-14 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Lung Diseases, Interstitial
Keywords: Interstitial lung disease; Scleroderma
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Diffuse | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Active Comparator): Tablet Tadalafil 20 mg every alternate day
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Tablet Placebo every alternate day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tab. Tadalafil 20 mg every other day for 6 months
  Arms: Tadalafil
Drug: Placebo — Shape , size, color and odor matched Tab. of inert material every other day for 6 months
  Arms: Placebo

SUMMARY:
Systemic sclerosis (SSc, scleroderma) is a multisystem autoimmune rheumatic disease that causes inﬂammation, vascular damage and ﬁbrosis. Besides involvement of skin, fibrosis also affects lung and heart. Although advances in understanding in pathophysiology and use of immunosuppressive therapy has brought significant improvement in outcome of other autoimmune diseases, scleroderma still remains as a disease with high mortality and 10 yr survival rate has improved only from 54% to 66% during last 25 years1. The frequency of deaths due to renal crisis significantly decreased (mainly due to effectiveness of ACE Inhibitors), from 42% to 6% of scleroderma-related deaths (p 0.001), whereas the proportion of patients with scleroderma who died of pulmonary fibrosis increased (due to lack of significant treatment) from 6% to 33% (p 0.001). However, presently, trials with immunosuppressive drugs including cyclophosphamide and other targeted molecules like Bosentan and Imatinib mesylate have shown very modest results at the best and given the risk of toxicity. The investigators have conducted three clinical trials with PDE5 inhibitor Tadalafil in the refractory Raynaud's phenomenon (RP) in SSc over last 3 years and had found good response in RP, healing of digital ulcers, prevention of new digital ulcers and also observed improvement in skin tightening, endothelial dysfunction and improvement of quality of life. The investigators therefore hypothesize that tadalafil may have an efficacy in improving the ILD of SSc.

The investigators therefore design this double-blind, randomized, placebo-controlled trial of oral Tadalafil (20 mg alternate day) in patients with SSc having ILD. Patients will be randomly assigned in a 1:1 ratio to receive either Tadalafil or matched placebo and will be followed up for 6 months. Prednisolone (if required for indications other than ILD) will be allowed up to 10 mg/d in all patients. Patient/s requiring more than 10 mg/d of prednisolone or equivalent dose of steroid will be excluded from the study. Patients who will fail on therapy during the study will be excluded from the study and will be asked to choose any therapeutic option from the rescue protocol.

Patients with FVC ≤ 70% predicted or DLCO ≤ 70 % of predicted, Evidence of ILD on HRCT will be enrolled. The primary objective of the study will be the change in FVC (expressed as a percentage of the predicted value) from baseline values at the end of 6-months of treatment. The secondary objectives will be improvement in dyspnea, improvement in 6 min walk distance, change in DLCO, change in total lung capacity, change in the disability index of the Health Assessment Questionnaire (S HAQ), and change quality of life (SF-36), levels of NT pro-BNP and fibrosis markers.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc, scleroderma) is a multisystem autoimmune rheumatic disease that causes inﬂammation, vascular damage and ﬁbrosis. Besides involvement of skin, fibrosis also affects many internal organ involving blood vessel, lungs, heart, kidney etc. Although advances in understanding in pathophysiology and use of immunosuppressive therapy has brought significant improvement in outcome of other autoimmune diseases, scleroderma still remains as a disease with high mortality and 10 yr survival rate has improved only from 54% to 66% during last 25 years1. But there is a significant change in pattern of cause of mortality over these years. The frequency of deaths due to renal crisis significantly decreased (mainly due to effectiveness of ACE Inhibitors), from 42% to 6% of scleroderma-related deaths (p 0.001), whereas the proportion of patients with scleroderma who died of pulmonary fibrosis increased (due to lack of significant treatment) from 6% to 33% (p 0.001). The frequency of pulmonary hypertension, independent of PF, also significantly increased during this time period (p<0.05)1. Presently PAH and interstitial lung disease accounts for majority of scleroderma related deaths. This emphasizes the need of novel therapies for interstitial lung disease in scleroderma, in order to improve the mortality and morbidity outcome of these patients.

The ﬁbrosis of the skin and internal organs in SSc is believed to be caused by the transition of quiescent ﬁbroblasts to activated myofibroblasts, which characteristically overproduce dermal ﬁbrillar collagen (type I, III, V), collagen-modifying enzymes and other extracellular matrix (ECM) components2. One of the major cytokines involved in this process is transforming growth factor TGF β1 3. TGF-β is normally secreted as a latent complex, which is required to be activated in extracellular regions before binding its receptors and exerting its biological effects. In dermal ﬁbroblasts, several membrane proteins, including integrin αVβ5 and thrombospondin 1(TSP1), catalyze the activation of latent TGF-β in the local microenvironment4,5. Binding of TGF-β to type II receptors (TRII) recruits type I receptors (TRI) and activates a series of signaling transduction pathways including the core Smad pathway (canonical pathway) and the non-Smad pathways (mitogen-activated protein kinase [MAPK], Rho, etc). TRI phosphorylates Smad3 at the S423/S425 within the C-terminal MH2. The activated pSmad3 binds with Smad4 to form the activated heteromeric Smad complex. The pSmad3/Smad4complexes enter the nucleus and associate with other transcription factors to regulate transcriptions of target genes required for collagen synthesis, myofibroblasts transformation and synthesis of matrix metalloproteinases6.

Studies of cyclophosphamide have shown inconsistent result on pulmonary function and survival. In the Scleroderma Lung Study (oral cyclophosphomide), there was only modest improvement in dyspnoea score, stabilization (no improvement) of FVC and no effect on DLCO at 1 year 7. At 2 years, there is no significant difference between any of these parameters between placebo and treatment group8. In a decision analysis using the Markov model to assess quality-adjusted life years (QALYs), authors conclude that there is no survival or quality of life benefit with oral cyclophosphamide9. Subsequent, Fibrosing Alveolitis in Scleroderma Trial (FAST) [intravenous cyclophosphamide followed by azathioprine] did not demonstrate significant improvement in the primary or secondary end points in the active treatment group versus the group receiving placebo10. A recent meta-analysis concluded that although previous trials with cyclophosphamide show a statistically significant improvement in lung function, they do not show a clinically significant improvement (>10% change in lung function)10. Considering the risk of infection and other serious adverse effects of oral cyclophosphamide, the risk benefit ratio may not be favorable for long term use of this drug. The experience with other immunosuppressive agents like mycophenolate moeftil11, azathioprine (as single agent)12,rituximab13 are limited to case studies or open label studies and lack double blind randomized control studies. Nonetheless, the potential adverse effects associated with these agents raise concern regarding their long term administration in a chronic disease like SSc -ILD.

Therefore, the focus of treatment of SSc associated ILD gradually shifting from non- specific immunosuppressive drugs to specific targeted therapy. Many attempts have been made to use drugs which target the molecular pathways responsible for causing fibrosis. Imatinib mesylate is a small molecule that blocks specific tyrosine kinases, including c-Abl and platelet-derived growth factor receptor (PDGFR) kinase. Incubation of cultured fibroblasts from patients with SSc and healthy volunteers with imatinib strongly inhibited the synthesis of col 1a1, col 1a2 and fibronectin-1 on the mRNA as well as protein level by up to 90% at concentrations of 1.0 mg/ml14. Treatment with imatinib completely prevented the development of fibrosis in the mouse model of Bleomycin-induced dermal fibrosis and tight-skin-1 (tsk-1) mouse model of SSc15. But clinical trials in patients failed to reproduce this effect. In a randomized, placebo-controlled trial of patients with mild to moderate Idiopathic pulmonary fibrosis followed for 96 weeks, imatinib did not affect survival or lung function16. The major adverse events include edema, muscle cramps and creatine kinase elevations, uncontrollable diarrhea and bone marrow toxicity, congestive heart failure17. These adverse effects need particular attention in clinical trials with patients with SSc because these patients often present with cardiac involvement, diarrhea and coexisting myositis with creatine kinase elevations. In addition, mild to moderate edema might be less well tolerated by patients with SSc with existing skin diseases than by patients with cancers 18.

Recently, endothelin1 (ET-1), is implicated in the pathophysiology of lung fibrosis. Endothelin 1(ET-1) is known to induce fibroblast chemotaxis and proliferation19, promote deposition of collagen20, decrease collagenase activity, and increase levels of fibronectin21. But Bosentan, a nonselective Endothelin receptor antagonist, in randomized placebo controlled trial failed to have any significant impact on 6-min walk distance or in lung function parameters 22.

PDE5 enzyme degrades cyclic guanosine monophosphate (c-GMP), a molecule responsible for nitric oxide-mediated vasodilatation. Recently PDE 5 inhibitors have shown to have novel antifibrotic effect by increasing level of CGMP. Cyclic GMP in turn activates the cGMP-dependent protein kinase G (PKG). Phosphorylation of Smad3 at S309 and T368 within MH2 by PKG prevents its heterodimerization with Smad4 and thus disrupts their nuclear translocation, resulting in repression of transcriptional activation23. TSP1 (thrombospondin -1) is a molecule catalyzing latent TGF-b activation and is expressed at high levels in cultured SSc ﬁbroblasts (in vitro) and in activated ﬁbroblasts in lesional skin of SSc (in vivo). Blockade of TSP1 by cyclic GMP partially abolishes the autocrine TGF-b signaling in SSc ﬁbroblasts24. Increase in level of cGMP blocks ca2+ pump and thereby improves endothelial disruption which is the initiating event in pathogenesis of fibrosis. Increase in NO level also helps in mopping up reactive oxygen species which are implicated in pathogenesis of fibrosis. In a Bleomycin induced pulmonary fibrosis model, PDE5 inhibition alters pulmonary and right ventricular (RV) response to intratracheal Bleomycin and that this inhibition acts through suppression of tissue free radicals and the Rho kinase pathway25. Dunkern et al showed that predominant PDE activities in lung fibroblasts are attributed to PDE5, PDE1 and to a smaller extent to PDE4 and PDE inhibitors prevent the formation of myofibroblasts from fibroblast 26.

The evidence that PDE 5 inhibitors are antifibrotic have mainly came from its effectiveness in prevention and treatment of Peyronie's disease (PD). In a rat model of TGF-β1-induced PD, Valente and associates, demonstrated that both oral sildenafil, a PDE5 inhibitor that protects cGMP from breakdown, and oral pentoxifylline, a predominantly PDE4 inhibitor that increases cAMP synthesis, counteract the development of the PD-like plaque27. In the case of pentoxifylline, it was proposed that the well-known cAMP-cGmP signaling crosstalk may be responsible for its antifibrotic effects. In a subsequent study in the same rat model, it was shown that another PDe5 inhibitor, vardenafil, given orally and in different dosing regimens, not only prevented but partially reversed the formation of the PD-like plaque. Preventive treatment at the higher dose reduced the overall collagen content, collagen iii/i ratio and the number of myofibroblasts and tGF-β1-positive cells, and selectively increased the apoptotic index of cells (presumably including myofibroblasts), in the PD-like plaque28. The antifibrotic effect although initially demonstrated in penile tissue, now proved in other tissues like heat, kidney and lungs. These antifibrotic effects of PDE5 inhibitors were also seen in rat models of diabetic nephropathy29, experimental glomerulonephritis24, myocardial infarction and hypertrophy30, and pulmonary fibrosis. So as scleroderma patients have fibrosis in multiple organs, the beneficial effect of PDE5 inhibitor may become manifold. It has also found to be very effective in treating other clinical manifestation of systemic sclerosis like PAH and digital ulcer. In a double-blind, randomized, placebo-controlled trial of sildenafil in idiopathic pulmonary fibrosis, there were significant differences in arterial oxygenation, carbon monoxide diffusion capacity, degree of dyspnea, and quality of life in patients treated with sildenafil in comparison to placebo group31. Tadalafil is a PDE5 inhibitor which is longer acting than sildenafil. It is safe and not associated with any serious life threatening side effect in the recently concluded study of effect of tadalafil in digital ulcer of scleroderma patients from our center32. In the same trial, Patients reported improvement of skin tightening and they can move their limb and joint more freely. Those patients with ILD had improvement or at least stabilization of lung function (Unpublished). Besides, FMD (flow mediated vasodilation as marker of endothelial dysfunction) significantly improved in these patients so providing another basis for using this drug for treatment of pulmonary fibrosis.

Hypothesis:

Tadalafil, a PDE5 inhibitor, by virtue of its stabilizing effect on endothelial dysfunction and anti-fibrotic effect, may have efficacy in reducing symptoms due to interstitial lung disease in scleroderma.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfillment of the criteria for systemic sclerosis (SSc) by American College or Rheumatology (ACR) criteria (Subcommittee for Scleroderma Criteria, 1980)
2. Forced vital capacity (FVC) ≤ 70% predicted.
3. DLCO ≤ 70 % of predicted

3. Presence of dyspnea on exertion (grade 2 on the Magnitude of Task component of the Mahler Modified Dyspnea Index) 4. Evidence of ILD on HRCT

Exclusion Criteria:

1. Those that cannot perform PFT or 6 min walk test
2. High dose prednisolone (1 mg/kg) or cyclophosphamide (> 500 mg) or MMF (> 500mg/d) or (azathioprine > 1 mg/kg) for more than 4 weeks anytime within previous 6 months
3. SBP < 90 mmHg or history of orthostatic hypotension
4. Current smokers
5. Women who are pregnant or lactating
6. Those receiving nitrates, alpha blockers, or both, other phosphodiesterase inhibitors
7. Current use of captopril (because of sulfhydryl group). If ACE- inhibitors are indicated, an ACE-inhibitor other than captopril should be used.
8. Serum creatinine ≥ 2.0 mg/dl.
9. Obstructive lung disease (FEV1/FVC ratio < 0.6)
10. Prostacyclins or endothelin antagonists or who had received any investigational drug within the prior month
11. Acute coronary or cerebrovascular event within 3 months
12. Evidence of malignancy
13. Peptic ulcer
14. Hepatic dysfunction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in FVC (expressed as a percentage of the predicted value) | 6 months
  To assess the change in FVC (expressed as a percentage of the predicted value) from baseline values at the end of 6 months

SECONDARY OUTCOMES:
Improvement in dyspnoea (as measured by Mehler dyspnoea index) | 6 months
  To assess the improvement in dyspnoea (as measured by Mehler dyspnoea index) at the end of 6 month
Improvement in 6 min walk test | 6 months
  To assess improvement in 6 min walk test at the end of 6 months
change in DLCO | 6 months
  To assess the change in DLCO from baseline values at the end of 6 months
change in total lung capacity | 6 months
  To assess the change in total lung capacity from baseline values at the end of 6 months
change in the disability index of the Health Assessment Questionnaire (S HAQ) | 6 months
  To assess the change in the disability index of the Health Assessment Questionnaire (S HAQ) at 6 months from baseline
change in the Medical Outcomes Study 36-item Short-Form General Health Survey (SF-36)scores | 6 months
  To assess the change in the Medical Outcomes Study 36-item Short-Form General Health Survey (SF-36) from baseline to end of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Agarwal, MD, DM, Principal Investigator — SGPGIMS
Locations (1):
- SGPGIMS, Lucknow, Uttar Pradesh, India